CLINICAL TRIAL: NCT05081700
Title: A Systems Approach to Understanding Disease Processes in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Providence Health & Services (Other)
Collaborators: Institute for Systems Biology (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ISB_PHS 2019-01
Record Dates: First submitted 2020-11-13; First posted 2021-10-18 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis
Keywords: multi-omic factors
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and stool samples will be analyzed for genetic and biochemical assay program including a whole genome sequence, advanced blood chemistry tests including heavy metals, proteins & metabolites, profiling of over 1000 low molecular weight metabolites and 29 fatty acids from blood plasma, measurement of nearly 200 serum proteins that constitute the neurology and inflammation panels of the O-link assay system, a description of the gut microbiome based on analysis of 16S ribosomal RNA sequences and serum immunoglobulin panel (IgG, IgM, and IgA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with relapsing MS: Patients with relapsing remitting MS who are intending to receive ocrelizumab.
  Interventions: Drug: All patients in the study will be treated with ocrelizumab

INTERVENTIONS:
Drug: All patients in the study will be treated with ocrelizumab — 300 mg of OCR IV infusion will be given on Day 0 followed by a second dose of 300 mg OCR 14 days later ± 2 days, and then 600 mg of OCR as a single infusion will be given every 24 weeks thereafter per standard medical care.
  Other Names: OCREVUS

SUMMARY:
This pilot study will establish a proof of concept for using a systems biology approach to characterize the dynamics of MS disease processes. The primary objective of the study is to identify multi-omic (genetic, proteomic, biochemical and/or microbial) factors that correlate with clinical and subclinical MS disease activity. Identification of such biomarkers could have an immediate clinical utility in identification of MS patients prone to more aggressive disease earlier in their disease course, thus affording the opportunity to better individualize therapy.

In addition, insights from better understanding of the complex interplay of various systems biology factors should improve our understanding of MS in general. The study will recruit 14 patients with relapsing MS who are initiating treatment with ocrelizumab, and follow them for 30 months.

DETAILED DESCRIPTION:
The main purpose of the study is to improve the understanding of MS and to look at the genetic factors that may influence how MS progresses. This will involve collecting blood and stool samples, patient questionnaires, and MS-related assessments.

About 67 mL (13 tsp) of blood will be collected at the first visit, and again at 6 months, 12 months, and 30 months after first visit.

Participants will receive standard treatment (ocrelizumab) and have standard exams, MRIs, and tests while on the study.

Study participation is about 30 months, which includes about 9 study visits. Some study visits may be up to 5 hours long. 14 people will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the purpose and risk of the study and provide written informed consent.
2. Male or female patients aged 18 to 60, inclusive at time of consent, who meet FDA approved indications to receive ocrelizumab treatment.
3. Have a definite diagnosis of relapsing MS (RMS) (Lublin et al. 2014).
4. Screening EDSS ≤ 5.0.
5. Have a length of disease duration since disease symptom onset ≤ 15 years.
6. Documentation of 1 or more on-DMT relapses, or 1 brain MRI revealing new or enlarged T2 lesion(s) over the 2 years prior to the screening visit (this could include DMT naïve patients).
7. Patient does not have any clinically significant medical conditions based on medical history, physical examination, and laboratory screening, as defined by the investigator, which would interfere with the conduct of the study.
8. Patient is willing and able to comply with the protocol assessments and visits, in the opinion of the investigator.
9. For women of childbearing potential: agreement to use an effective birth control method and avoid breastfeeding during the study period, and for those patients who have received ocrelizumab, for at least 6 months after the last dose.

Inclusion criteria for those patients who have completed the core study and are re-consenting and re-enrolling to complete the month 30 visit. Patients must fulfill all of the following criteria to participate in the study:

1. Able to understand the purpose and risk of the study and provide written informed consent.
2. Have participated in the core study and continue to receive ocrelizumab.
3. Have not passed week 120±14 days post initial ocrelizumab dose in the core study.
4. Diagnosis of relapsing MS at time of consent.
5. Patient is willing and able to comply with the protocol assessments and visits, in the opinion of the investigator.
6. For women of childbearing potential: agreement to use an effective birth control method and avoid breastfeeding during the study period and for at least 6 months after the last dose of ocrelizumab.

Exclusion Criteria:

1. Diagnosis of progressive MS at screening.
2. Patient is unable to undergo MRI with gadolinium contrast imaging for any reason.
3. Known presence of other neurological disorders, including but not limited to, the following:

   1. History of cerebrovascular disorders.
   2. History or known presence of CNS tumor.
   3. History or known presence of potential metabolic causes of myelopathy.
   4. History of peripheral neuropathy.
   5. History or known presence of infectious disease of the CNS.
   6. History of genetically inherited CNS degenerative disorder.
   7. Neuromyelitis optica spectrum disorder, anti-Aquaporin 4 IgG, or Anti-MOG IgG .
   8. History of progressive multifocal leukoencephalopathy (PML).
   9. History or known presence of any other concurrent systemic or nervous system autoimmune disorders, potentially causing progressive neurologic disease.
   10. History of severe, clinically significant brain or spinal cord trauma (e.g., cerebral contusion, spinal cord compression).
4. Exclusions related to general health:

   1. Pregnancy or lactation.
   2. Chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study.
   3. History or currently active primary or secondary immunodeficiency.
   4. Lack of peripheral venous access.
   5. Hypersensitivity to ocrelizumab or to any of its excipients.
   6. Significant or uncontrolled non-neurological systemic disease.
   7. Significant active infections must be treated and resolved before possible inclusion in the study.
   8. Patients in an immunocompromised state.
   9. Patients with history of malignancy, except for adequately treated basal cell skin cancer or in situ cervical cancer.
5. Exclusions Related to Medications:

   1. Your last COVID-19 vaccine should be given at least 2 weeks before and all vaccines should be given at least 6 weeks before the first infusion of ocrelizumab. Live/live attenuated vaccines should be avoided during treatment and safety follow-up period until B cells are peripherally repleted to at least the lower limit of normal. COVID-19 vaccines are permitted per investigator discretion during ocrelizumab treatment.
   2. Treatment with any investigational agent within 24 weeks of screening (Visit 1) or five half-lives of the investigational drug (whichever is longer) or treatment with any experimental procedures for MS (e.g., treatment for chronic cerebrospinal venous insufficiency) within 24 weeks of screening (Visit 1).
   3. Previous treatment with B-cell targeted therapies (i.e., rituximab, ocrelizumab, atacicept, tabalumab, belimumab, ofatumumab, or obinutuzumab).
   4. Any previous treatment with total body irradiation, or bone marrow transplantation.
   5. Previous treatment with natalizumab in the past 4 weeks prior to baseline (Day 0) or fingolimod in the last 2 weeks prior to screening (Visit 1).
   6. Patients previously treated with teriflunomide, unless an accelerated elimination procedure is implemented and/or teriflunomide serum level of less than 2 mcg/ml is documented prior to screening (Visit 1).
   7. Previous treatment with azathioprine, mycophenolate mofetil or methotrexate in the last 12 weeks prior to screening (Visit 1).
   8. Previous treatment with cyclosporine or cladribine at any time in the past in the last 96 weeks prior to screening (Visit 1).
   9. Previous treatment with mitoxantrone, alemtuzumab, or cyclophosphamide at any time.
   10. Treatment with dalfampridine unless on stable dose for ≥30 days prior to screening (Visit 1). Wherever possible, patients should remain on stable doses throughout the treatment period.
6. Exclusions related to laboratory findings:

   1. Positive serum β-human chorionic gonadotropin (hCG) measured at screening.
   2. Positive screening tests for hepatitis B (hepatitis B surface antigen [HbsAg] positive, or positive hepatitis B core antibody [total HbcAb], or other comparable tests confirmed by a positive viral DNA polymerase chain reaction [PCR]), within the 6 months prior to Day 0.
   3. Positive tuberculin skin test or Quantiferon Gold TB test, unless previously documented treatment for latent TB within the 12 months prior to Day 0 or a negative test within the 12 months prior to Day 0.
   4. Evidence of acute or chronic hepatitis, or evidence of clinically significantly impaired hepatic function through clinical and laboratory evaluation including alkaline phosphatase >1.5x ULN, ALT or AST >2x ULN; GGT>3x ULN or bilirubin >ULN.
   5. Any other clinically significant laboratory abnormality which may put the patient at risk.

Exclusion criteria for those patients who have completed the core study and are re-consenting and re-enrolling to complete the month 30 visit. Patients must be excluded from participating in the study if they meet any of the following criteria:

1. Exclusions related to general health:

   1. Pregnancy or lactation.
   2. Chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study.
2. Exclusions Related to Medications:

   1. Live/live attenuated vaccines should be avoided during treatment and safety follow-up period until B cells are peripherally repleted to at least the lower limit of normal. COVID-19 vaccines are permitted per investigator discretion during ocrelizumab treatment.
   2. Treatment with dalfampridine unless on stable dose. Wherever possible, patients should remain on stable doses throughout the treatment period.
3. Exclusions related to laboratory findings:

   1. Any clinically significant laboratory abnormality during the study which may put the patient at risk.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Study patients will be recruited from the population of relapsing MS patients initiating treatment with ocrelizumab, who are being followed at the Swedish MS Center in Seattle, Washington and the Providence MS Center in Portland, Oregon.
  MS population and a reference non-MS population
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Proportion of relapse free patients | 6, 12, and 30 months
  Number of participants free of MS relapse at 6, 12, and 30 months divided by total number of participants.

SECONDARY OUTCOMES:
Annualized relapse rate (ARR) | 12 and 30 months
  Changes in ARR to assess MS activity levels at baseline compared to 12 and 30 months. Total number of relapses divided by total number of participants.
Correlates of T2 lesions on-study MRI activity | 12, 24, and 30 months
  Number of new and/or unique T2 lesions for each participant compared to screening
Correlates of gadolinium enhancing lesions on-study MRI activity | 12, 24, and 30 months
  Number of new and/or enlarged gadolinium enhancing lesions for each participant compared to screening
Expanded Disability Status Scale (EDSS) | 12 and 30 months
  Changes in EDSS to assess MS activity levels at baseline compared to 12 and 30 months. The EDSS provides a total score on a scale that ranges from minimum 0 to maximum 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability
Timed 25-Foot Walk (T25FW) | 6, 12, and 30 months
  Changes in T25FW to assess MS activity levels at baseline compared to 6, 12, and 30 months. Scale ranges from minimum 0 seconds to maximum 180 seconds. Lower score indicates better result.
9-Hole Peg Test (9HPT) | 6, 12, and 30 months
  Changes in 9HPT to assess MS activity levels at baseline compared to 6, 12, and 30 months. Scales ranges from minumum 0 seconds to maximum 300 seconds (5 minutes). Lower score indicates better result.
Low Contrast Visual Acuity (LCVA) | 6, 12, and 30 months
  Changes in LCVA to assess MS activity levels at baseline compared to 6, 12, and 30 months. Test performed on right eye, left eye, and binocular (both eyes). Scale ranges from minimum 20/200 to maximum 20/16. Higher score indicates better result.
Symbol digit modality test (SDMT) | 6, 12, and 30 months
  Changes in SDMT to assess MS activity levels at baseline compared to 6, 12, and 30 months. Scale ranges from minimum 0 to maximum 110. Higher score indicates better result.
Modified Fatigue Impact Scale (MFIS) | 6, 12, and 30 months
  Changes in MFIS to assess MS activity levels at baseline compared to 6, 12, and 30 months. Scale ranges from minimum 0 to maximum 84. Lower score indicates better result.
Beck Depression Inventory (BDI-2) | 6, 12, and 30 months
  Changes in BDI-2 to assess MS activity levels at baseline compared to 6, 12, and 30 months. Scale ranges from minimum 0 to maximum 63. Lower score indicates better result.

OTHER OUTCOMES:
Whole genome sequencing | 6, 12, and 30 months
  Exploratory use of advanced blood chemistry including 3072 proteomic, 930 lipidomic, 1348 metabolite, and thousands of microbiome feature profiles in patients with multiple sclerosis to determine if these measures provide valid biomarkers for assessing prognosis and response to therapy.
Blood analysis plasma | 6, 12, and 30 months
  Exploratory profiling of over 1000 low molecular weight metabolites and 29 fatty acids from blood plasma to determine if these measures provide valid biomarkers for assessing prognosis and response to therapy.
Blood analysis serum | 6, 12, and 30 months
  Measurement of approximately 3,072 serum proteins that constitute the neurology, neuro-exploratory and inflammation panels of the O-link assay system, and/or global plasma protein analysis (O-Link Explore 3072).
Extracellular vesicle analysis plasma | 6, 12, and 30 months
  An in-depth proteomic analysis of extracellular vesicles from blood plasma. This is a potential refinement of the proteomic data already obtained by isolation of extracellular vesicles and subjecting them to comprehensive proteomic analysis.
Stool analysis gut microbiome | 12 and 30 months
  Description of the gut microbiome based on analysis of shotgun sequencing from stool samples.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Cohan, MD, PhD, Principal Investigator — Providence Health & Services
Locations (2):
- United States (2):
  - Providence Neurological Specialties West, Portland, Oregon
  - Swedish Medical Center Multiple Sclerosis Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
It is expected that the results of this study will be presented at the annual meetings of American Academy of Neurology (AAN) and European Committee for Treatment and Research in Multiple Sclerosis (ECTRIMS). In addition, a manuscript reporting the results of this study will be submitted for publication in a leading neurology journal in aggregate, no intention to disclose individual personal data.

REFERENCES:
- [Background] Ontaneda D, Thompson AJ, Fox RJ, Cohen JA. Progressive multiple sclerosis: prospects for disease therapy, repair, and restoration of function. Lancet. 2017 Apr 1;389(10076):1357-1366. doi: 10.1016/S0140-6736(16)31320-4. Epub 2016 Nov 24. PMID 27889191
- [Background] Steinman L, Zamvil SS. Beginning of the end of two-stage theory purporting that inflammation then degeneration explains pathogenesis of progressive multiple sclerosis. Curr Opin Neurol. 2016 Jun;29(3):340-4. doi: 10.1097/WCO.0000000000000317. PMID 27027554
- [Background] Fraussen J, de Bock L, Somers V. B cells and antibodies in progressive multiple sclerosis: Contribution to neurodegeneration and progression. Autoimmun Rev. 2016 Sep;15(9):896-9. doi: 10.1016/j.autrev.2016.07.008. Epub 2016 Jul 7. PMID 27396817
- [Background] Price ND, Magis AT, Earls JC, Glusman G, Levy R, Lausted C, McDonald DT, Kusebauch U, Moss CL, Zhou Y, Qin S, Moritz RL, Brogaard K, Omenn GS, Lovejoy JC, Hood L. A wellness study of 108 individuals using personal, dense, dynamic data clouds. Nat Biotechnol. 2017 Aug;35(8):747-756. doi: 10.1038/nbt.3870. Epub 2017 Jul 17. PMID 28714965
- [Background] Hellberg S, Eklund D, Gawel DR, Kopsen M, Zhang H, Nestor CE, Kockum I, Olsson T, Skogh T, Kastbom A, Sjowall C, Vrethem M, Hakansson I, Benson M, Jenmalm MC, Gustafsson M, Ernerudh J. Dynamic Response Genes in CD4+ T Cells Reveal a Network of Interactive Proteins that Classifies Disease Activity in Multiple Sclerosis. Cell Rep. 2016 Sep 13;16(11):2928-2939. doi: 10.1016/j.celrep.2016.08.036. PMID 27626663
- [Background] Hakansson I, Tisell A, Cassel P, Blennow K, Zetterberg H, Lundberg P, Dahle C, Vrethem M, Ernerudh J. Neurofilament light chain in cerebrospinal fluid and prediction of disease activity in clinically isolated syndrome and relapsing-remitting multiple sclerosis. Eur J Neurol. 2017 May;24(5):703-712. doi: 10.1111/ene.13274. Epub 2017 Mar 6. PMID 28261960
- [Background] Cekanaviciute E, Yoo BB, Runia TF, Debelius JW, Singh S, Nelson CA, Kanner R, Bencosme Y, Lee YK, Hauser SL, Crabtree-Hartman E, Sand IK, Gacias M, Zhu Y, Casaccia P, Cree BAC, Knight R, Mazmanian SK, Baranzini SE. Gut bacteria from multiple sclerosis patients modulate human T cells and exacerbate symptoms in mouse models. Proc Natl Acad Sci U S A. 2017 Oct 3;114(40):10713-10718. doi: 10.1073/pnas.1711235114. Epub 2017 Sep 11. PMID 28893978